CLINICAL TRIAL: NCT03952182
Title: Effect of Bracing Versus No Bracing in Stable Thoracolumbar Compression and Burst Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and follow up concerns during Covid-19 pandemic
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, William Behrens, MD, Resident Physician, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29976
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Thoracic Fracture; Lumbar Fracture; Compression Fracture of Thoracic Vertebral Body; Compression Fracture of Lumbar Spine; Burst Fracture of Thoracic Vertebra; Burst Fracture of Lumbar Vertebra
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Orthosis (LSO, TLSO, etc) (Active Comparator): Patient's in this arm will be given an orthosis for the treatment of their injury (TLSO for thoracic or upper lumbar injury, LSO for lumbar injury)
  Interventions: Other: Spinal Orthosis (LSO, TLSO)
- No Spinal Orthosis (Experimental): the patient's in this arm will not be given an orthotic. They will be given a bending restriction and otherwise remain activities as tolerated.
  Interventions: Other: No orthosis

INTERVENTIONS:
Other: Spinal Orthosis (LSO, TLSO) — spinal orthosis prescribed for specific spinal fracture (TLSO for thoracic or high lumbar fracture, LSO for lumbar fracture)
  Arms: Spinal Orthosis (LSO, TLSO, etc)
Other: No orthosis — no orthotic given for spinal fracture. These patient's will be given a bending restriction
  Arms: No Spinal Orthosis

SUMMARY:
Spinal orthoses have been used in the treatment of non-operative thoracic and lumbar fractures with much success. However, there has been increasing questioning as to wether or not the orthotics are necessary to have a good overall outcome. Being fitted for and acquiring braces are associated with great expense and increased hospital stays. The purpose of this study is to determine wether or not braces are required for good outcome post thoracic or lumbar fracture.

DETAILED DESCRIPTION:
Several tens of patient's per year come to the Emergency Department with thoracolumbar spine compression and burst fractures that are not indicated for surgical fixation. Currently, these patients are treated non-operatively through brace wear which is either custom made for the patient or is off-the-shelf pending location of the fracture and surgeon preference. All braces are through the currently contracted orthotics company. As they are non stocked in house, waiting for the brace requires the patients to remain on "strict spine precautions" (flat bed rest in a Miami J collar, no pillows behind the head, and logrolls for turning) for anywhere from 24-48 hours. No only is this incredibly uncomfortable for the patient, it is also extending their hospital stay for at least one day and, sometimes, up to three as they wait for the brace and have it adjusted to fit appropriately. The patient's all have to then wait to work with physical therapy and occupational therapy and, finally, have upright spine films taken in the brace. The braces tend to be very uncomfortably and constricting for patient's and significantly inhibit their daily lives. The investigators are proposing that these fractures can be treated without needing bracewear and will have equivalent to superior outcomes than results while wearing the brace.

ELIGIBILITY:
Inclusion Criteria:

* Any acute, stable thoracic or lumbar compression or burst fracture appropriate for non-operative care

Exclusion Criteria:

* neurological deficit, pregnant, incarcerated, non-English speaking, previous spinal surgery, additional lower extremity injury affecting weight bearing, younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 6 month post-injury
  Primary outcome is the ODI which is a a self-completed questionnaire over ten topics regarding pain, lifting, ability to perform activities of daily living, ability to walk, sit, stand, one's sexual function, social life, sleep quality, and ability to travel. Each category has six different statements from which the patient can choose to best describe their current status. Each question is then scored on a scale from 0-5. Scores are summed and then doubled. The index is from 0-100 with zero being no disability and one hundred being maximally disabled.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Time of injury and at follow up at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  VAS is a continuous scale represented as a horizontal line with vertical dashes numbered 0-10. Each number is given a pain intensity descriptor that ranges from "no pain" (score of 1) to "worst imaginable pain" (score of 10). The patient is asked to rate the pain they are currently experiencing on that scale from 1-10
SF-12 | time of injury and follow up at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
PROMIS (Patient-Reported Outcomes Measurement Information System)- physical function | time of injury and follow up at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  PROMIS is a U.S. NIH initiative that is an item bank of self-administered questions to measure physical function. This includes functionality of one's upper extremities (dexterity), lower extremities (mobility), neck, back, as well as ability to perform activities of daily living. This assessment measures current function rather than function over a time period. Each question has five response options ranging in value from 1-5. The total raw score for the form is the sum of the values of the response to each question. The raw score (which can range from 10 (worst) to 50 (best) is then compared to a PROMIS specific conversion chart to the appropriate T-score. A T-score of roughly 50 is considered 'average' and 'slightly sicker than the general population'.
Return to Work Status | follow up at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Patient's will be asked if they currently work at time of injury and at each consecutive follow up appointment will be asked if they have returned to work

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University Hospital, St Louis, Missouri, United States